CLINICAL TRIAL: NCT02175082
Title: A Forced Cycling Exercise Program in Individuals With Parkinson's Disease: Can it Improve Gait Parameters?
Brief Title: Cycling in Parkinson's Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated prior to enrollment goals due to difficulty with recruiting subjects
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Northwestern Memorial Hospital (Other); Paul Ruby Foundation for Parkinson's Research (Unknown)
Responsible Party: Principal Investigator, Christina Marciniak, Professor, Northwestern University and Attending Physician, Shirley Ryan AbilityLab, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00093757
Record Dates: First submitted 2014-06-21; First posted 2014-06-26 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinson Disease; Exercise; Rehabilitation; Physical Therapy; Cycling
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: Subjects were randomized to a delay start or immediate start group and then for the cycling, the intervention was randomized to : forced pace (80-90 revolutions per minute with equals 15 miles per hour cycling rate or self-selected with both groups working at similar aerobic levels
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and those performing outcome assessments were not aware of group allotment, nor was the PI. The therapists supervising the exercise interventions were aware of the group allotment
Oversight: Data Monitoring Committee: No

ARMS (2):
- Forced exercise cycling (Active Comparator): Cycling exercise at approximately 90 rpm
  Interventions: Other: Cycling at Forced rate
- Self-selected pace cycling (Active Comparator): Cycling at self selected rate, with same aerobic level as forced cycling group
  Interventions: Other: Cycling at self-selected rate

INTERVENTIONS:
Other: Cycling at Forced rate
  Arms: Forced exercise cycling
Other: Cycling at self-selected rate
  Arms: Self-selected pace cycling

SUMMARY:
The purpose of this study is to assess the effectiveness of a forced exercise aerobic exercise program, utilizing a cycling activity, on specific gait parameters and balance in individuals with Parkinson's Disease (PD). Design: pilot, feasibility, randomized control, evaluator blinded. Subjects: Twenty four patients with idiopathic PD Hoehn and Yahr (H&Y) stage II or III. Intervention: Participants randomly assigned to one of two exercise groups, forced exercise or self selected exercise, on cycling machine three times a week for 8 weeks. Both groups to exercise at same aerobic intensity level to keep heart rate at 60-80% heart rate max. Outcomes: Gait parameters of step length, width, and variability as measured by the GAITRite; 6 Minute Walk Test; mini-BESTest (balance testing); exercise tolerance via Patient Reported Outcomes Measurement Information System (PROMIS) scale.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's Disease
* Hoehn and Yahr Stages II - III.
* Ages 30-80 years
* Medical Clearance
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* MOCA: (Montreal Cognition Scale) : rating of less than 24, indicative of cognitive dysfunction
* Changes in Parkinson's medications within the two weeks prior to starting the study
* Anticipated change in Parkinson Disease medications during the course of the study
* Uncontrolled orthostasis
* Symptomatic coronary artery disease
* Fracture of lower limb within 6 months prior to study onset or significant lower limb orthopedic diagnosis that would limit cycling
* Other significant neurologic diagnoses including multiple sclerosis or vestibular disease
* Acute illness
* Physical therapy within the month prior to study entry
* Subjects already participating in a forced exercise or high intensity exercise program
* Any medical condition that the physician investigator determined would compromise safety.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
6-minute walk test | 8 weeks
  Distance walked in 6 minutes

SECONDARY OUTCOMES:
Stride length | 8 weeks
  Length of stride in meters as measured by the GAITrite
Step Width | 8 weeks
  Width of step in meters as measured by the GAITrite
Step variability | 8 weeks
  Standard deviation of step as measure in meters by the Gaitrite system
10 meter walk test | 8 weeks
  Time in seconds for the subject to walk 10 meters
miniBESTest (Balance Evaluation Systems Test) | 8 weeks
  Subject is scored as the 14 activities on this scale are performed, and a summary score is derived.

OTHER OUTCOMES:
Steps per day | Over 8 week trial and for 2 months post intervention
  Subjects steps per day will be measured with a Garmin wrist step counter

CONTACTS AND LOCATIONS:
Overall Officials: Christina M Marciniak, MD, Principal Investigator — Shirley Ryan AbilityLab/Northwestern University Chicago IL
Locations (1):
- Shirley Ryan AbilityLab (formerly the Rehabilitation Institute of Chicago), Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sung P, Rafferty M, Doyle L, Kliver E, Bines K, Traines J, Scarpa A, Marciniak C, Solanki S, Todd A. Technology-based Forced Paced Cycling in Parkinson's disease: Is it Feasible and Effective?Archives of PM&R October 2019Volume 100, Issue 10, Page e126
- See also: Meeting abstract published — https://doi.org/10.1016/j.apmr.2019.08.377